CLINICAL TRIAL: NCT03639207
Title: IFNL4 Genotype for Predicting Response to Ledipasvir/Sofosbuvir: Kaiser Permanente Northern California
Brief Title: IFNL4 Genotype for Predicting Response to Ledipasvir/Sofosbuvir
Status: Withdrawn | Type: Observational
Why Stopped: Subject Research)
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999918134; 18-C-N134
Record Dates: First submitted 2018-08-18; First posted 2018-08-21 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis C Virus
Keywords: IFNL4; Genetics; Ledipasvir/Sofosbuvir Treatment
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients treated with ledipasvir/sofosbuvir in the Kaiser Permanente Northern California

SUMMARY:
Background:

Hepatitis C virus (HCV) infection is a leading cause of hepatocellular carcinoma and end-stage liver disease. Ledipasvir/sofosbuvir is used to treat chronic HCV. The drug name for it is Harvoni. It is a very effective treatment, but it is expensive. Researchers have found a genetic variation that predicts how people will respond to this treatment. They want to learn more about this genetic link. It could help develop better treatments for HCV.

Objective:

To study if certain inherited genetic differences and other factors affect the different ways patients respond to treatment with Harvoni.

Eligibility:

Adults ages 18 who are members of the Kaiser Health Plan and have recently been treated for hepatitis C with Harvoni

Design:

Researchers will review medical records to identify a group of people who could be in the study.

Participants will provide a saliva sample at home. They will get instructions and kit to collect it in.

Participants will spit into a funnel until it reaches a mark on the funnel. It will be about 1 teaspoon of saliva with no bubbles.

They will return the sample in a prepaid mailer.

Researchers will do genetic tests on the samples. The participant data will be kept confidential. It will not be given to insurance companies.

Participants will not be given any test results.

...

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is a leading cause of hepatocellular carcinoma (HCC) and end stage liver disease - successful treatment markedly reduces those risks. Ledipasvir/sofosbuvir is a highly effective, but expensive, treatment for chronic hepatitis C. Previously, we demonstrated that genetic variation in IFNL4 predicts response to this regimen. We now propose to examine the association between genotype for the functional IFNL4-DeltaG/TT polymorphism and treatment response among patients enrolled in a large managed care organization. In a two-stage design, limited demographic and clinical data for patients who have been treated with ledipasvir/sofosbuvir will be ascertained from an electronic database. In the second stage, additional demographic and clinical data will be extracted from medical records and consented patients will provide a specimen for IFNL4 genotyping. These data will be combined to examine associations of IFNL4-DeltaG/TT genotype and other variables with response to ledipasvir/sofosbuvir. We will also develop a clinical prediction model for response to ledipasvir/sofosbuvir treatment. These results could inform more efficient treatment of HCV in the United States and globally.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subject Inclusion Criteria:

* At least 18 years of age
* Chronic HCV VGT-1 infection
* Completed treatment with ledipasvir/sofosbuvir (with or without ribavirin) for either 8, 12 or 24 weeks at a participating KP-NC clinical site
* Data available to determine virological relapse and SVR12

EXCLUSION CRITERIA:

Subject Exclusion Criteria:

* Otherwise eligible subjects who have left KPNC will not be included in the study
* Otherwise eligible subjects who cannot provide informed consent in English will not be included in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with ledipasvir/sofosbuvir in the Kaiser Permanente Northern California
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-06-15 (Estimated); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
IFNL4-deltaG/TT polymorphism and treatment response to ledipasvir/sofosbuvir | 12 weeks post treatment
  virological relapse

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R O'Brien, M.D., Principal Investigator — National Cancer Institute (NCI)